CLINICAL TRIAL: NCT00460395
Title: Surgery Versus Stereotactic Radiosurgery in the Treatment of Single Brain Metastasis: A Randomized Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NS97-199
Record Dates: First submitted 2007-04-12; First posted 2007-04-16 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Brain Cancer
Keywords: Brain Metastasis; Cerebral Metastases; Brain Cancer; Stereotactic Radiosurgery; Craniotomy
MeSH Terms: conditions — Brain Neoplasms | interventions — Surgical Procedures, Operative; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Surgery
Procedure: Stereotactic radiosurgery

SUMMARY:
Study Objectives:

* To compare the survival (overall, systemic, and neurological) of patients with single cerebral metastases treated with either conventional surgical resection or stereotactic radiosurgery.
* To compare their rates of recurrence, complications, and their cognitive ability, functional status, and quality of life.

Although surgical resection is a proven and effective treatment for brain metastases in patients with systemic cancer, stereotactic radiosurgery has been suggested to be equally effective and less morbid. Nonrandomized retrospective comparisons have been unable to resolve whether stereotactic radiosurgery is as effective as conventional surgery because of the complexity and variability of the population of patients with cancer and brain metastases. This controversy can only be resolved by a prospective randomized trial comparing these treatment modalities. Patients not randomized will be analyzed as a separate group.

DETAILED DESCRIPTION:
Eligible patients will be randomized to either conventional surgery or stereotactic radiosurgery, or participate as a separate group of the study, if they refuse randomization. At the time of diagnosis, patients may be given dexamethasone which will be continued throughout treatment then discontinued in a tapered fashion. Patients with supratentorial tumors and a history of seizures may be treated with anticonvulsants. For patients in the surgical group, surgery will be performed using standard techniques and any necessary intraoperative adjuncts. For patients in the stereotactic radiosurgery group, stereotactic radiosurgery will be delivered using the modified linear accelerator and multiple non-coplanar converging arcs. The dose prescribed will be dependent on the volume treated. Changes in patients' clinical courses will be treated as medically necessary. Should metastases recur or progress at the primary intracerebral site or at a distant intracerebral site, patients who received radiosurgery remain eligible for surgical resection and patients who received conventional surgery may undergo repeat resection or radiosurgery. Whole brain radiotherapy may be given to patients who demonstrate local or distant recurrence and can be given as the primary therapy or as adjunctive therapy. The WBRT dose will be 30 Gy delivered in ten fractions.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years and older;
* Documented diagnosis of cancer within 5 years (except for patients with unknown primary);
* Newly diagnosed single brain metastases as determined by MRI;
* Candidacy for both conventional surgical resection as well as stereotactic radiosurgery;
* Karnofsky Performance Score > 70;
* Life expectancy of at least 4 months;
* Signature of the approved consent form.

Exclusion Criteria:

* Prior radiation therapy to the brain;
* Evidence of leptomeningeal disease;
* Need for immediate treatment to prevent neurological deterioration;
* Extremely radiosensitive primary tumor;
* Prior radioiodine (for thyroid metastases);
* Pregnancy or lactation.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 1998-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick F. Lang, M.D., Principal Investigator — Universtity Of Texas MD Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org